CLINICAL TRIAL: NCT03045991
Title: The Effects and Mechanism of the Sequential Combination of Exercise and Cognitive Training on Cognitive Function in Stroke Patients With Cognitive Decline: A Randomized Controlled Trial
Brief Title: Effects and Mechanism of the Sequential Combination of Exercise and Cognitive Training in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201600871A3
Record Dates: First submitted 2016-12-12; First posted 2017-02-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stroke Patients With Cognitive Decline
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential training group (SEQ) (Experimental): The sequential training group (SEQ) will first receive 30-minutes aerobic exercise training followed by 30-minutes computerized cognitive training. All participants will receive a training session for 60 minutes per day, three days per week for 12 weeks, a total of 36 training sessions.
  Before and after the treatment, a total of 2 evaluations were conducted, including clinical assessments and blood test (each 18c.c.). A saliva sample (2 mL) will only be collected once from each subject. A follow-up assessment of clinical outcomes will be conducted at six month after the end of the course of treatment.
  Interventions: Behavioral: aerobic exercise training; Behavioral: cognitive training
- control intervention group (CI) (Active Comparator): The control intervention group (CI) will receive a control training session for 60 minutes per day, three days per week for 12 weeks, a total of 36 training sessions.
  Before and after the treatment, a total of 2 evaluations were conducted, including clinical assessments and blood test (each 18c.c.). A saliva sample (2 mL) will only be collected once from each subject. A follow-up assessment of clinical outcomes will be conducted at six month after the end of the course of treatment.
  Interventions: Behavioral: control training

INTERVENTIONS:
Behavioral: aerobic exercise training — The aerobic exercise program using progressive resistive stationary bicycle training which will contain warm-up, resistive physical exercise, and cool-down. The training resistance will increase with improvement of participants' performance.
  Arms: sequential training group (SEQ)
Behavioral: control training — The control training program will receive 30 minutes non-aerobic exercise training, including stretching muscle skills, joint mobility exercises; in addition to one 30-minute session of unstructured mental activities, such as reading books or reading educational films.
  Arms: control intervention group (CI)
Behavioral: cognitive training — The computerized cognitive training program will be implemented with the brainHQ to target abilities of visuospatial processing, attention, memory, and executive function. The level of the training program will become more difficult with progress in participants' targeted cognitive abilities.
  Arms: sequential training group (SEQ)

SUMMARY:
The purpose of this study is to determine the treatment effects of sequential combination of aerobic exercise and cognitive training on cognitive function, physiological markers, daily function, physical function, social participation and quality of life in stroke patients with cognitive decline.

DETAILED DESCRIPTION:
Cognitive decline after stroke is a common sequela and is highly associated with functional disability. Empirical evidence shows that exercise combined cognitive training may induce neuroplastic changes that modulate cognitive function. However, evidence about the effects of combined exercise-cognitive trainings on physiological biomarkers, cognitive and physical functions in stroke patients with cognitive decline is still less. The present study aim to investigate the effects of sequential combination of exercise-cognitive trainings on cognitive, physical, and daily function. In addition, the physiological mechanism of the combination training on cognitive function by several biomarkers including the brain-derived neurotrophic factor (BDNF), antioxidative marker, HbA1c, and plasma lipid level will be investigated. This study is a single-blind randomized controlled trial. Participants will be randomly assigned to SEQ group in which sequentially perform physical exercise and cognitive training or to CI group of control intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke occurring at least 6 months prior to enrollment
2. MMSE score ≥ 19,MoCA<26,able to follow the study instruction
3. Self- or informant-reported memory or cognitive complaints or CDR scale ≤ 0.5
4. Adequate cardiopulmonary function to perform aerobic exercise
5. Able to walk with or without assistive devices

Exclusion Criteria:

1. Unstable medical history (e.g., recent myocardial infarction) that might limit participation
2. Concomitant with other neurological disorders (e.g., Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis)
3. Current participation in another interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09; Primary Completion 2019-10-16 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The MoCA will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30
Change scores of Wechsler Memory Scale - Third Edition (WMS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The WMS-III is a standardized and reliable neuropsychological examination tool designed to evaluate visuospatial and memory functions
Change scores of Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The WAIS-III is developed to measure an individual's intelligence level. It includes tests that evaluate cognitive functions in verbal comprehension, working memory, perceptual organization, and processing speed
Change scores of Useful Field of View (UFOV) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The UFOV assessment is a computer-based visual test containing three subtests: visuomotor processing speed, divided attention, and selective attention.
Change scores of Stroop Color-Word test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Stroop Color-Word assesses the abilities of selective attention, inhibition and executive function. The participants will be tested under congruent and incongruent conditions.
Change scores of Dual-task test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The dual-task test evaluates the ability to shift attention between one task and another. Participants will perform the box and block test (BBT) while doing secondary cognitive tasks while sitting. Participants will perform BBT by affected and less affected hand.

SECONDARY OUTCOMES:
Change scores of serum BDNF level | Baseline, posttest (an expected average of 3 months)
  Up-regulation of neurotrophic and vascular growth factors
Change scores of Antioxidative marker | Baseline, posttest (an expected average of 3 months)
  Antioxidative markers will be used to reflect the changes on oxidative stress. In particular, we will be analyzing the total antioxidant capacity (TAC).
Change scores of Glucose indicator | Baseline, posttest (an expected average of 3 months)
  HbA1C level will be tested to investigate the relationships between blood glucose level and aerobic exercise
Change scores of Plasma lipid level | Baseline, posttest (an expected average of 3 months)
  The cholesterol ratio (total cholesterol divided by high-density lipid) will be evaluated to reflect the lipid level in the blood.
Change scores of Functional Independence Measure (FIM) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The FIM assesses the dependence level of individuals with stroke to perform 18 activities (13 motor and five cognitive tasks) in daily living. The score ranges from 18 to 126 and higher scores demonstrate greater independent participation in daily activities.
Change scores of Lawton Instrumental Activities of Daily Living Scale (Lawton IADL) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Lawton IADL scale assesses independent living skills, such as shopping or managing finances.
Change scores of Stroke Impact Scale (SIS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The SIS 3.0 will be used to evaluate health-related quality of life for patients with stroke. The SIS assesses eight domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function) with 59 test items.
Change scores of Caregiver Burden (CB) scale | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  CB scale evaluates the burden of the primary caregiver of the participants. Lessening the burden of caregivers after the intervention may significantly improve the quality of life for patients with stroke and their family.
Change scores of EuroQol (EQ)-5D questionnaire | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The quality of life will be assessed by the EQ-5D questionnaire which comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change scores of Timed up and go test (TUG) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down.
Change scores of Six-minute walk test (6MWT) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The 6MWT measures the maximum distance walked over 6 minutes, which assess the endurance and mobility level of the participants. The participants could rest as needed during the course of the test.
Change scores of Mobility level | Baseline, posttest (an expected average of 3 months)
  Accelerometers will be used to provide an objective measure of the amount of arm movements in real-life situations. The participants will be asked to wear an Actigraphy activity monitor.
Change scores of International Physical Activity Questionnaires (IPAQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The IPAQ is an international measure of health-related physical activity.
Change scores of Fugl-Meyer Assessment (FMA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The UE-FMA subscale will be used to assess the sensorimotor impairment level of UE in patients after stroke. The UE-FMA contains 33 movements with a score range from 0 to 66. A higher UE-FMA score indicates less impairment of the paretic limb. The validity and reliability of FMA is good to excellent.
Change scores of Rivermead Mobility Index (RMI) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The RMI evaluates the participant's bed mobility, postural transfers and walking ability. It contains a 15-item scale which includes 14 questions and one direct observation, with a total of score of 15.
Change scores of muscle strength | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Accelerometers will be used to provide an objective measure of the amount of arm movements in real-life situations. The participants will be asked to wear an Actigraphy activity monitor.
  We will evaluate isometric knee flexors and extensors muscle strength using handheld dynamometer. Also, we will use hand dynamometer to measure grip strength of the affected and less affected hand while the participant is seated, with the elbow at 90-degree flexion. We will record the mean value of 3 attempts.
Change scores of Community Integration Questionnaire (CIQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The CIQ measures items relevant to home integration, social integration, and productive activities.
Change scores of Geriatric Depression Scale (GDS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Chinese version of short form GDS will be used.
Genotyping of the BDNF val66met polymorphism | Once during the intervention(an expected average of 3 months)
  Up-regulation of neurotrophic and vascular growth factors
Change scores of Actigraphy | Baseline, posttest (an expected average of 3 months)
  In addition to MAL, the ActiGraph GX3 accelerometers (ActiGraph, Shalimar, FL, USA) will be used to quantitatively assess the amount of arm use in the participants' home settings.The actigraphy will be placed on bilateral wrist for 3 consecutive days before and after the 1-month intervention. The participants will carry the actigraphy all day except for activities that involve water, such as swimming or bathing. Using the actigraphy, investigators will be able to record and calculate the number of hand movements per minute, and the data will be analyzed with the MAHUFFE software (http://www.mrc-epid.cam.ac.uk/). The actigraphy has often been used to evaluate arm use in patients with stroke.
Change scores of Mini-Mental State Exam (MMSE) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of Medical Research Council scale (MRC) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The MRC is an ordinal scale that assesses muscle strength. The scoring for each muscle ranges from 0 to 5, with a higher score indicates stronger muscle. The reliability of MRC for all muscle groups was good to excellent in patients with stroke.
Change scores of National Institutes of Health Stroke Scale | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung University
Locations (6):
- Taiwan (6):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Keeling Chang Gung Memorial Hospital, Keelung
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Yeh TT, Chang KC, Wu CY. The Active Ingredient of Cognitive Restoration: A Multicenter Randomized Controlled Trial of Sequential Combination of Aerobic Exercise and Computer-Based Cognitive Training in Stroke Survivors With Cognitive Decline. Arch Phys Med Rehabil. 2019 May;100(5):821-827. doi: 10.1016/j.apmr.2018.12.020. Epub 2019 Jan 9. PMID 30639273